CLINICAL TRIAL: NCT02024035
Title: Health Economic Evaluation of Tomotherapy and Dynamic Arctherapy in ENT Epidermoid Carcinoma
Brief Title: Protocole Advanced RadioTherapy ORL
Acronym: ART-ORL
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Collaborators: The Biostatistics and Therapy Evaluation Unit (Other)
Responsible Party: Sponsor
Other Study IDs: ART-ORL; ET 2009-044
Record Dates: First submitted 2011-08-16; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Tomotherapy; Head and neck squamous celle carcinoma; Health economic evaluation
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Tomotherapy
  Interventions: Radiation: Radiotherapy
- Arc'therapy Vmat
  Interventions: Radiation: Radiotherapy
- Arctherapy Rapid'Arc
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy

SUMMARY:
The purpose of this study is to do health economic evaluation of tomotherapy and dynamic arctherapy (2 techniques exist: RapidArc and Vmat).

This study evaluate also local disease control after 18 months in patients with an ENT epidermoid carcinoma and treated by tomotherapy orarctherapy .

The number of patients required in this study is: 300:

* Number of patients treated with tomotherapy: 120
* Number of patients treated with dynamic arctherapy RapidArc: 120
* Number of patients treated with dynamic arctherapy Vmat: 60

This is a prospective; multicentric and non randomized study.

ELIGIBILITY:
Inclusion Criteria:

* PS <= 2
* Age >= 18 years
* Histologically proven carcinoma
* Cavum Epidermoïd or undifferentiated carcinoma; or oropharynx epidermoïd carcinoma; or oral cavity epidermoïd carcinoma
* Stade T1 to T4
* M0
* Patient with no surgery ( except laser partial surgery and ganglionic cleaning out)
* Bilateral ganlionic cervical area irradiation
* Covered by a medical insurance.

Exclusion Criteria:

* Prior history of other malignancies in the last 5 years(except non evolutive ENT cancer or squamous cell carcinoma )
* Re-irradiation indication
* Unilateral cervical area irradiation
* Post-operative radiotherapy
* Patient treated by amifostine
* Impossible follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Cavum Epidermoïd or undifferentiated carcinoma; or oropharynx epidermoïd carcinoma; or oral cavity epidermoïd carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2009-11; Primary Completion 2012-03 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The various of cost between tomotherapy and Intensity Modulation Radiation Therapy (IMRT) | 18 months
  The purpose of this study is to realise a Health economic evaluation of the various cost between tomotherapy and Intensity Modulation Radiation Therapy (IMRT)

SECONDARY OUTCOMES:
The economic impact of the learning curve of the tomotherapy process, the operating procedures and the activity of the centres | 18 months
  To estimate the economic impact of the learning curve of the tomotherapy process, the operating procedures and the activity of the centres
To determine the difference of cost for the preparation phase and the irradiation phase of the radiotherapy procedure | 18 months
  One of the secondary objectives for the economic evaluation is to individualize the difference of cost for the preparation phase and the irradiation phase of the radiotherapy procedure
The salivary toxicity | at 6; 12 and 18 months post treatment
  The salivary function will be assessed at baeline; 6; 12 and 18 months post treatment.
  This evaluation will be done with differents scale (RTOG, EVA); and with salivary scan.
To determine the rate of disease local control | Baseline, Month 6; Month 18
  Assement of disease by clinical exam and/or imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe GIRAUD, PhD, Principal Investigator — Hopital Europeen Georges Pompidou, Paris; FRANCE
Locations (14):
- France (14):
  - Institut Sainte Catherine, Avignon
  - Institut BERGONIE, Bordeaux
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Centre Privé de Radiothérapie de Metz, Metz
  - Centre Val d'Aurelle, Montpellier
  - Centre Alexis Vautrin, Nancy
  - Intitut Curie, Paris
  - Hôpital Eurppéen Geoges POMPIDOU, Paris
  - Centre Eugène Marquis, Rennes
  - Centre René GAUDUCHEAU, Saint-Herblain
  - Centre Paul STRAUSS, Strasbourg
  - Groupe Oncorad Garonne, Toulouse
  - Institut Claudius Regaud, Toulouse

REFERENCES:
- [Derived] Bibault JE, Dussart S, Pommier P, Morelle M, Huguet M, Boisselier P, Coche-Dequeant B, Alfonsi M, Bardet E, Rives M, Calugaru V, Chajon E, Noel G, Mecellem H, Servagi Vernat S, Perrier L, Giraud P. Clinical Outcomes of Several IMRT Techniques for Patients With Head and Neck Cancer: A Propensity Score-Weighted Analysis. Int J Radiat Oncol Biol Phys. 2017 Nov 15;99(4):929-937. doi: 10.1016/j.ijrobp.2017.06.2456. Epub 2017 Jun 27. PMID 28864403
- [Derived] Bibault JE, Morelle M, Perrier L, Pommier P, Boisselier P, Coche-Dequeant B, Gallocher O, Alfonsi M, Bardet E, Rives M, Calugaru V, Chajon E, Noel G, Mecellem H, Perol D, Dussart S, Giraud P. Toxicity and efficacy of cetuximab associated with several modalities of IMRT for locally advanced head and neck cancer. Cancer Radiother. 2016 Jul;20(5):357-61. doi: 10.1016/j.canrad.2016.05.009. Epub 2016 Jun 23. PMID 27345843